CLINICAL TRIAL: NCT00008827
Title: The Use of the Internet to Facilitate Weight Loss and Maintenance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: HarveyBerinoInternet (cmpltd); R01DK056746 (NIH)
Record Dates: First submitted 2001-01-17; First posted 2001-01-17 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: Obesity; Behavioral weight control; Internet
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Behavioral: Behavioral weight loss

SUMMARY:
This project is assessing the effectiveness of using the Internet as a tool to facilitate the maintenance of weight lost in a behavioral weight control program. Participants attend a standard behavioral weight control intervention via Interactive Television and after 6 months are randomly assigned to one of three groups; a control group, an in-person weight maintenance group and a maintenance group that meets over the Internet. This research project is being conducted in Vermont.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 39.9
* Internet connection

Exclusion Criteria:

* Major medical problems
* Inability to walk for exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Jean Harvey-Berino, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States